CLINICAL TRIAL: NCT01028391
Title: A 30-Week Extension to: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of the Initial Therapy With Coadministration of Sitagliptin and Pioglitazone in Patients With Type 2 Diabetes Mellitus
Brief Title: 30-Week Extension to an Initial Combination Study (24 Weeks in Duration) of Sitagliptin With Pioglitazone (0431-064)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-064-10; MK0431-064-10; 2009_003
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin + Pioglitazone (Experimental)
  Interventions: Drug: Sitagliptin 100 mg q.d.+ Pioglitazone 45 mg q.d.; Drug: Metformin
- Pioglitazone + Placebo (Active Comparator)
  Interventions: Drug: Pioglitazone 45 mg q.d. + Sitagliptin 100 mg placebo q.d.; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin 100 mg q.d.+ Pioglitazone 45 mg q.d. — Patients will receive combination therapy with blinded sitagliptin 100 mg q.d. (q.d. = once daily) and open-label pioglitazone 45 mg q.d. during the up to 30 week extension study. Sitagliptin 100 mg q.d. and pioglitazone 45 mg q.d. will be administered as oral tablets.
  Arms: Sitagliptin + Pioglitazone
Drug: Pioglitazone 45 mg q.d. + Sitagliptin 100 mg placebo q.d. — Patients will receive placebo to match sitagliptin 100 mg q.d. (blinded) and open-label pioglitazone 45 mg q.d. during the up to 30 week extension study. The placebo to match sitagliptin 100 mg q.d. (blinded) and open-label pioglitazone 45 mg q.d. will be administered as oral tablets.
  Arms: Pioglitazone + Placebo
Drug: Metformin — Patients not meeting specific glycemic goals during the 30-week extension study will receive open-label metformin at a dose determined by the investigator.

SUMMARY:
A 30-week extension to a 24-week study assessing the hemoglobin A1c (HbA1c)- and fasting plasma glucose (FPG)-lowering efficacy of the combination of sitagliptin and pioglitazone in patients with type 2 diabetes mellitus (T2DM) with inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Patients must complete the double-blind base study (MK-0431-064-00)(NCT00397631) and have at least 75% compliance with study medication during the base study treatment period.
* Women of childbearing potential must continue to comply with the protocol-specified contraceptive methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yoon KH, Shockey GR, Teng R, Golm GT, Thakkar PR, Meehan AG, Williams-Herman DE, Kaufman KD, Amatruda JM, Steinberg H. Effect of initial combination therapy with sitagliptin, a dipeptidyl peptidase-4 inhibitor, and pioglitazone on glycemic control and measures of beta-cell function in patients with type 2 diabetes. Int J Clin Pract. 2011 Feb;65(2):154-64. doi: 10.1111/j.1742-1241.2010.02589.x. PMID 21235696
- [Derived] Yoon KH, Steinberg H, Teng R, Golm GT, Lee M, O'Neill EA, Kaufman KD, Goldstein BJ. Efficacy and safety of initial combination therapy with sitagliptin and pioglitazone in patients with type 2 diabetes: a 54-week study. Diabetes Obes Metab. 2012 Aug;14(8):745-52. doi: 10.1111/j.1463-1326.2012.01594.x. Epub 2012 Apr 17. PMID 22405352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in the 30-week extension study: 21-Sep-2007.
  Last patient last visit of the 30-week extension
  study: 23-Jan-2009; 53 study centers worldwide.
Pre-assignment Details: Patients ≥18 years with type 2 diabetes mellitus (T2DM) and hemoglobin A1c (HbA1c) of 8-12% on diet/exercise meeting all other entry criteria were eligible for participation in the 24-week base study.
  Patients who completed the base study with >75% study drug compliance were eligible to enter the 30-week extension study at participating sites.
Groups:
- Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d.: The Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. (q.d. = once daily) group includes extension study data from patients who received once-daily coadministered treatment with oral tablets of sitagliptin 100 mg and pioglitazone 45 mg. During the 24-week base study (prior to the entering the extension study), these patients received once-daily coadministered treatment with oral tablets of sitagliptin 100 mg and pioglitazone 30 mg.
- Pioglitazone 45 mg q.d.: The Pioglitazone 45 mg q.d. (q.d. = once daily) group includes extension study data from patients who received once-daily coadministered treatment with oral tablets of placebo to sitagliptin 100 mg and pioglitazone 45 mg. During the 24-week base study (prior to entering the extension study), these patients received once-daily coadministered treatment with oral tablets of placebo to sitagliptin 100 mg and pioglitazone 30 mg.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. | Pioglitazone 45 mg q.d.
Started | 164 | 153
Completed | 150 | 142
Not Completed | 14 | 11
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 3 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Needed excluded medication | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. | Pioglitazone 45 mg q.d. | Total
Number analyzed (Participants) | 164 | 153 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] — These data reflect the patients' ages at the beginning of the 24-week base study
  years | 51.4 (10.0) | 52.3 (11.5) | 51.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 63 | 141
  Male | 86 | 90 | 176
Race/Ethnicity, Customized [Number; unit: participants]
  White | 93 | 85 | 178
  Black | 7 | 3 | 10
  Asian | 42 | 41 | 83
  Other | 22 | 24 | 46
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] — These data reflect the baseline measurement at the beginning of the 24-
  week base study. The number of patients with data for HbA1c at this time point were N=163 (sitagliptin+pioglitazone),
  N=151 (pioglitazone), and N=314 (total).
  Percent | 9.4 (1.2) | 9.4 (1.2) | 9.4 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (i.e., Week 0 of the 24-week Base Study) in Hemoglobin A1c (HbA1c) at Week 54
Description: HbA1c is measured as percent. Thus this change from baseline reflects the Week 54 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and 54 Weeks
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 value for this outcome during the 30-week extension study. For FAS patients with no data at Week 54, the last observed measurement during the 30-week extension study was carried forward to Week 54.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent HbA1c
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. | Pioglitazone 45 mg q.d.
Number analyzed (Participants) | 161 | 149
Percent HbA1c | -2.37 [-2.54 to -2.19] | -1.86 [-2.04 to -1.68]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. vs Pioglitazone 45 mg q.d; Test type: Superiority or Other; Mean Difference (Net) = -0.51, 95% CI [-0.76 to -0.26], Standard Error of Mean 4.0 — This is a difference in least squares means, based on an ANCOVA model with terms for treatment and baseline (i.e., Week 0 of the 24-week base study) HbA1c

2. Secondary Outcome: Change From Baseline (i.e., Week 0 of the 24-week Base Study) in Fasting Plasma Glucose (FPG) at Week 54
Description: Change from baseline at Week 54 is defined as Week 54 minus Week 0.
Time Frame: Baseline and Week 54
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 value for this outcome during the extension study. For FAS patients with no data at Week 54, the last observed measurement during extension study was carried forward to Week 54.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. | Pioglitazone 45 mg q.d.
Number analyzed (Participants) | 163 | 152
mg/dL | -61.3 [-66.7 to -55.9] | -52.8 [-58.4 to -47.2]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. vs Pioglitazone 45 mg q.d; Test type: Superiority or Other; Mean Difference (Net) = -8.5, 95% CI [-16.3 to -0.7], Standard Error of Mean 4.0 — This is a difference in least squares means, based on an ANCOVA model with terms for treatment and baseline (i.e., Week 0 of the 24-week base study) FPG

ADVERSE EVENTS:
Time Frame: Weeks 24 to 54 (i.e., the entire 30-week extension study)
Description: Non-serious adverse experience results represent those events included in the prespecified primary analysis of safety (i.e., excluding events that occurred following the initiation of glycemic rescue therapy) for this study.
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. | Pioglitazone 45 mg q.d.
Serious Adverse Events (participants affected / at risk) | 5/164 | 3/153
Other Adverse Events (participants affected / at risk) | 8/164 | 8/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. (N=164) | Pioglitazone 45 mg q.d. (N=153)
All Cardiac Disorders (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
All Infections and Infestations (Infections and infestations) | 3 | 2
Appendicitis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1
All Nervous System Disorders (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg q.d. + Pioglitazone 45 mg q.d. (N=164) | Pioglitazone 45 mg q.d. (N=153)
All Infections and Infestations (Infections and infestations) | 8 | 8
Nasopharyngitis (Infections and infestations) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.